CLINICAL TRIAL: NCT00129571
Title: A Phase 1 Dose Escalation Study of the Safety and Pharmacokinetics of XL820 Administered Orally to Subjects With Solid Tumors
Brief Title: Study of XL820 in Adults With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Exelixis (Industry)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: XL820-001
Record Dates: First submitted 2005-08-10; First posted 2005-08-12 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-06

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

INTERVENTIONS:
Drug: XL820

SUMMARY:
The purpose of this study is to assess the safety and tolerability of XL820 when given orally to adults with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Advanced solid tumor
* Cancer for which standard therapies do not exist or are no longer effective
* Life expectancy of > 3 months
* Adequate bone marrow, liver, and kidney function
* Willing to use accepted method of contraception during the course of the study
* Negative pregnancy test (females)
* Written informed consent

Exclusion Criteria:

* Chemotherapy within 4-6 weeks of the start of treatment (depending on the therapy)
* Radiotherapy to more than 25% of bone marrow within 4 weeks of the start of treatment
* Investigational drug within 30 days of the start of treatment
* Subjects with known brain metastasis
* Uncontrolled medical disorder such as infection or cardiovascular disease
* Subjects known to be HIV positive
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-08

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Cancer Therapy and Research Center, San Antonio, Texas